CLINICAL TRIAL: NCT05169853
Title: Correlation Between Programmed Death-Ligand1 Expression and Clinical Outcomes After Neoadjuvant Systemic Therapy in Her-2 Positive and Triple Negative Breast Cancer
Brief Title: Programmed Death-Ligand1 Expression in Her-2 Positive and Triple Negative Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Akram, Principle Investigator, Ain Shams University
Other Study IDs: MD 177/2021
Record Dates: First submitted 2021-11-24; First posted 2021-12-27 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Triple Negative Breast Cancer; HER2-positive Breast Cancer
Keywords: breast cancer; her-2 positive; triple negative; neoadjuvant therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Patients with Her-2 positive and triple negative breast cancer who received neoadjuvant chemotherapy will be included in the study. Paraffin blocks of preoperative core or tru-cut biopsies of the participants will be collected and tested for programmed death-ligand 1 (PD-L1) expression. The variation of PD-L1 expression among different breast cancer subtypes will be evaluated and the investigator will correlate between PD-L1 expression and pathological complete response to neoadjuvant systemic therapy.

DETAILED DESCRIPTION:
Files of breast cancer patients attending breast cancer clinic at Ain Shams University Clinical oncology and nuclear medicine department will be viewed by the investigator and those who fit the selection criteria will be included in the study. Tru-cut or core tissue biopsies obtained from the participants for initial diagnosis will be collected and PD-L1 testing will be done on the specimens. Scoring of PD-L1 will be done using Combined positive score (CPS) score. PD-L1 expression will be evaluated among Her-2 positive and triple negative subtypes and will be correlated with pathological complete response after reviewing the postoperative pathology results of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or more
* Histologically proven invasive breast cancer
* Any T stage, any N Stage with no distant metastasis M0 as evident by clinical examination and sonomammography.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2.
* Patients with Her-2 positive Luminal B subtype, Her-2 enriched or triple negative breast cancer.
* Patients who completed their systemic neoadjuvant therapy.

Exclusion Criteria:

* Second malignancy
* Patients with early breast cancer clinicallyT1 (≤ 2 cm) N0
* Metastatic patients M1
* Patients with autoimmune diseases (Type I Diabetes mellitus, Systemic Lupus Erythematosus, Rheumatoid Arthritis, Sjogren's syndrome and Behcet disease)
* Patients on systemic steroids or other immunomodulators (as Methotrexate, Tacrolimus and Cyclosporine)
* Patients who started but didn't complete neoadjuvant systemic therapy
* Patients who didn't undergo surgery after neoadjuvant systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast Cancer patients attending Ain Shams University Clinical Oncology and Nuclear Medicine Department breast clinic from 2016 till 2021 with the following selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Variation of PD-L1 expression in Her-2 positive and triple negative breast cancer | through study completion, an average of 1 year
  We will compare between percentage of PD-L1 positive cases in the studied Her-2 positive and triple negative breast cancer subtypes
Correlation between pathological complete response and PD-L1 expression | through study completion, an average of 1 year
  We will correlate between PD-L1 expression and pathological complete response in the studied cases

CONTACTS AND LOCATIONS:
Overall Officials: Iman A Sharawy, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Clinical Oncology Department, Cairo, Abbasseya, Egypt